CLINICAL TRIAL: NCT03007004
Title: Trial to Confirm the Effect and Safety of Local Injection of Botulinum Toxin Type B Against Digital Ulcer in Systemic Sclerosis
Brief Title: Effect and Safety of Local Injection of Botulinum Toxin Type B Against Digital Ulcer in Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gunma University (Other)
Responsible Party: Principal Investigator, Sei-ichiro Motegi, Associate Professor, Gunma University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2016017
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Systemic Sclerosis Patients With Digital Ulcers
Keywords: Systemic aclerosis; digital ulcer; botulinum toxin
MeSH Terms: conditions — digital ulcers | interventions — rimabotulinumtoxinB; batrachotoxinin A 20-alpha-benzoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Botulinum toxin group (Experimental): 400 units in one injection site（0.2mL） Total 2000 units（1.0mL） （For both hands total 4000 units; 2.0 mL）
  Interventions: Drug: Botulinum toxin type B (2500 units / vial)
- Physiological saline (control drug) group (Sham Comparator): 0.2mL in one injection site
  Total 1.0mL (For both hands total 2.0 mL)
  Interventions: Drug: Physiological saline

INTERVENTIONS:
Drug: Botulinum toxin type B (2500 units / vial) — BTX-B (E2014, Eisai, NerBloc®) was injected subcutaneously from the palmar side into seven locations around interphalangeal metacarpophalangeal joints, targeting the neurovascular bundles just proximal to the A1 pulley (the radial and ulnar sides of the first finger, the radial side of second finger, the ulnar side of the fifth finger and between the second to fifth fingers). Three locations between the second and third fingers, the third and fourth fingers, and the fourth and fifth fingers were injected with 400 U (0.2 ml) of BTX-B. In addition, the radial and ulnar sides of the first finger, the radial side of the second finger, and the ulnar side of the fifth finger were injected with half a dose of BTX-B (200 units; 0.1 ml). A total of 2000 U (1.0 ml) of BTX-B was injected into one hand. Injections were performed using a 30-gauge needle.
  Other Names: BTX-B (E2014, Eisai, NerBloc®)
  Arms: Botulinum toxin group
Drug: Physiological saline — Saline solution was injected subcutaneously from the palmar side into seven locations around interphalangeal metacarpophalangeal joints, targeting the neurovascular bundles just proximal to the A1 pulley (the radial and ulnar sides of the first finger, the radial side of second finger, the ulnar side of the fifth finger and between the second to fifth fingers). Three locations between the second and third fingers, the third and fourth fingers, and the fourth and fifth fingers were injected with saline (0.2 ml). In addition, the radial and ulnar sides of the first finger, the radial side of the second finger, and the ulnar side of the fifth finger were injected with half a dose of saline (0.1 ml). A total of 1.0 ml of saline was injected into one hand. Injections were performed using a 30-gauge needle.
  Arms: Physiological saline (control drug) group

SUMMARY:
Efficacy and safety of local infusion of botulinum toxin type B in patients with systemic sclerosis (SSc) with digital ulcer is evaluated by a randomized, double-blind study.

DETAILED DESCRIPTION:
To assess the efficacy and safety of local injection of botulinum toxin type B (BTX-B) against digital ulcers (DUs) and Raynaud's phenomenon (RP) in patients with systemic sclerosis (SSc).

In a randomized, double-blind, placebo-controlled, investigator-initiated clinical trial (phase II), 10 patients with SSc and RP-related DUs were randomly and evenly assigned to a placebo control group or treatment group taking BTX-B injections. The degree of improvement in DU, change in size, number of new DUs, improvement in symptoms of RP, and adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with SSc in diagnostic criteria (Appendix 1) by the American-European Rheumatology Association
2. Patients who have Raynaud's phenomenon from consultation, inquiries, etc. judged by Clinical responsibility (sharing) doctor
3. Patients with digital ulcer at acquiring consent The criteria for digital ulcers are as follows.

   * It is a peripheral ulcer from the proximal interphalangeal joint and the thumb interphalangeal joint (including the interphalangeal joint).
   * The continuity of coating by the epithelium has been lost and there is a depth that is visible to the eye. Incidentally, when exposed, cases covered with eschar or necrotic tissue are also included.
   * If the exposure is not clearly recognized (crusted or covered with necrotic tissue), the investigational responsibility (shared) doctor can judge that the epidermis and the dermis are missing.
   * It should not be the paronychia、crack、digital pitting scars.
   * It should not be attached to the projection of the calcification.
   * Size: The maximum diameter (major axis) is 0.5 cm or more.
   * Bones, tendons and joints are not exposed.
   * It is not accompanied by obvious infection findings.
4. At the time of acquiring consent Patients over 18 years old
5. Patients for whom consent has been obtained in writing on participation of this trial

Exclusion Criteria:

1. Patients with Raynaud's phenomenon due to diseases other than SSc
2. Patients with systemic neuromuscular junction disorder (myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis etc.)
3. Patients with advanced respiratory dysfunction
4. Patients with a history of hypersensitivity to components of botulinum toxin type B (botulinum toxin type B, human serum albumin, succinate buffer) or other botulinum toxin
5. Patients who received botulinum toxin formulation within 4 months before study drug administration or who have continued efficacy of botulinum toxin at the time of administration of investigational drug even when administered more than 4 months ago
6. Patients who received endothelin receptor antagonist within 60 days before study drug administration
7. Patients who received the following medications within 14 days prior to study drug administration

   * Argatroban hydrate injection
   * Prostaglandin E1 Injection (eg alprostadil injection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who completely lost index ulcer 8 weeks after administration | 8 weeks after administration
  The primary end point was the percentage of subjects with complete disappearance of index ulcer 8 weeks after administration. The index ulcer was defined as the largest DUs in the hand. The size of DU was measured as both the longest diameter of the ulcer and the diameter perpendicular to the center of the ulcer's diameter. Complete disappearance is defined as the disappearance of the area of the ulcer that has become epithelialized and covered by the epidermis from the periphery of the ulcer and continued coverage of the ulcer surface area that has been restored.

SECONDARY OUTCOMES:
the percentage of subjects with complete disappearance of index ulcer at 4, 12, and 16 weeks after administration | at 4, 12, and 16 weeks after administration
  the percentage of subjects with complete disappearance of index ulcer at 4, 12, and 16 weeks after administration
the rate of change in the number of DUs per hand | at 4, 8, 12, and 16 weeks after administration
  the rate of change in the number of DUs per hand
the number of newly formed DUs | at 4, 8, 12, and 16 weeks after administration
  the number of newly formed DUs
the number of newly formed DUs per hand | at 4, 8, 12, and 16 weeks after administration
  the number of newly formed DUs per hand
the changes in RP severity were assessed using Raynaud's Condition Score [RCS] | at 4, 8, 12, and 16 weeks after administration
  the changes in RP severity were assessed using Raynaud's Condition Score [RCS]. RCS is a daily self-assessment of RP activity using a 0-10 ordinal scale. RCS incorporates the cumulative daily frequency, duration, severity, and effect of RP attacks. RCS was averaged over a 7-day period preceding the baseline and each subsequent visit.
the changes of investigator rating Raynaud's Condition Score [RCS] | at 4, 8, 12, and 16 weeks after administration
  the changes of investigator rating Raynaud's Condition Score [RCS]. Investigator rating RCS was also assessed by the investigator (SM).
the changes in the score of pain/numbness severity assessed using the 100-mm Visual Analog Scale (VAS) | at 4, 8, 12, and 16 weeks after administration
  Pain/numbness severity was assessed using the 100-mm Visual Analog Scale (VAS). Pain/numbness severity was assessed using the 100-mm Visual Analog Scale (VAS) (range 0-100; 0 refers to no pain/numbness, and 100 refers to worst imaginable pain/numbness)
the changes of the recovery of skin temperature in the finger with the index ulcer | at 4, 8, 12, and 16 weeks after administration
  the skin temperature of the finger was measured just after and 10 minutes after an ice-bath immersion
the changes in the attack duration of Raynaud's phenomenon | at 4, 8, 12, and 16 weeks after administration
  the changes in the attack duration of Raynaud's phenomenon
the changes in the number of attacks of Raynaud's phenomenon per day | at 4, 8, 12, and 16 weeks after administration
  the number of attacks of Raynaud's phenomenon per day was assessed for 7days

CONTACTS AND LOCATIONS:
Overall Officials: Sei-ichiro Motegi, Principal Investigator — Gunma University
Locations (1):
- Gunma University Graduate school of Medicine, Morishita, Gunma, Japan